CLINICAL TRIAL: NCT04522167
Title: A Phase 3 Randomized, Double-masked, Multicenter Study to Compare the Efficacy and Safety of the Proposed Aflibercept FYB203 Biosimilar in Comparison to Eylea® in Patients With Neovascular Age-Related Macular Degeneration
Brief Title: Efficacy and Safety of the Aflibercept FYB203 Biosimilar in Comparison to Eylea® in Patients With Neovascular Age-Related Macular Degeneration
Acronym: MAGELLAN-AMD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bioeq GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FYB203-03-01
Record Dates: First submitted 2020-08-11; First posted 2020-08-21 (Actual); Results first posted 2025-11-13 (Actual); Last update posted 2025-11-13 (Actual); Status verified 2024-10

CONDITIONS: Neovascular Age-related Macular Degeneration
MeSH Terms: interventions — aflibercept

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- FYB203 (Proposed aflibercept biosimilar) (Experimental): Patients will receive intravitreal (IVT) injections of FYB203 as detailed in the protocol.
  Interventions: Drug: FYB203 (Proposed aflibercept biosimilar)
- Eylea® (Aflibercept) (Active Comparator): Patients will receive intravitreal (IVT) injections of Eylea® as detailed in the protocol.
  Interventions: Drug: Eylea® (Aflibercept)

INTERVENTIONS:
Drug: FYB203 (Proposed aflibercept biosimilar) — Patients will receive 1 IVT injection of FYB203 in the study eye only every 4 weeks for the first 3 consecutive doses, followed by 1 IVT injection every 8 weeks through study completion.
  Arms: FYB203 (Proposed aflibercept biosimilar)
Drug: Eylea® (Aflibercept) — Patients will receive 1 IVT injection of Eylea® in the study eye only every 4 weeks for the first 3 consecutive doses, followed by 1 IVT injection every 8 weeks through study completion.
  Arms: Eylea® (Aflibercept)

SUMMARY:
This is a randomized, double-masked, multicenter study to evaluate the efficacy and safety of FYB203 compared to Eylea® in patients with neovascular age related macular degeneration.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 50 years at Screening.
* Male or female:

  * Male: A male patient must agree to use contraception as defined in this protocol during the treatment period and for at least 4 weeks after the last dose of study treatment.
  * Female: A female patient is eligible to participate if she is not pregnant, not breastfeeding, and at least 1 of the following conditions applies:

    1. Not a woman of childbearing potential (WOCBP), OR
    2. A WOCBP who agrees to follow the contraceptive guidance during the treatment period and for at least 4 weeks after the last dose of study treatment.
* Capable of giving signed informed consent, which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.
* Willingness and ability to undertake all scheduled visits and assessments.
* Newly diagnosed choroidal neovascularization (CNV) lesion secondary to wet AMD

Exclusion Criteria:

Patients are not eligible for the study if any of the following criteria apply:

* Employees of clinical study sites, individuals directly involved with the conduct of the study or immediate family members thereof, prisoners, and persons who are legally institutionalized.
* Study eye requiring immediate treatment.
* Any prior treatment with VEGF agent or any investigational products to treat AMD in either eye.
* Uncontrolled ocular hypertension or glaucoma in the SE (defined as intraocular pressure [IOP] ≥ 30 mmHg, despite treatment with anti-glaucomatous medication).
* Ocular disorders in the SE (i.e. retinal detachment, pre-retinal membrane of the macula or cataract with significant impact on VA) at the time of screening that may confound interpretation of study results and compromise VA.
* Any concurrent intraocular condition in the SE (e.g. glaucoma, cataract, or diabetic retinopathy) that, in the opinion of the Investigator, would either require surgical intervention during the study to prevent or treat visual loss that might result from that condition or affect interpretation of study results.
* Use of other investigational drugs (excluding vitamins, minerals) within 30 days or 5 half lives from randomization, whichever is longer.
* Any type of advanced, severe, or unstable disease, including any medical condition (controlled or uncontrolled) that could be expected to progress, recur, or change to such an extent that it may bias the assessment of the clinical status of the patient to a significant degree or put the patient at special risk.
* Stroke or myocardial infarction within 6 months prior to randomization.
* Known hypersensitivity to the IMP (aflibercept or any component of the aflibercept formulation) or to drugs of similar chemical class or to fluorescein or any other component of fluorescein formulation.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 434 (Actual)
Dates: Start 2020-07-21 (Actual); Primary Completion 2022-06-23 (Actual); Study Completion 2023-05-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Official, Study Director — Bioeq GmbH
Locations (66):
- Bulgaria (2):
  - Research Site, Sofia
  - Research Site, Stara Zagora
- Czechia (5):
  - Research Site, Hradec Králové
  - Research Site, Ostrava
  - Research Site, Pardubice
  - Research Site, Prague
  - Research Site, Sokolov
- Hungary (7):
  - Research Site, Budapest
  - Research Site, Debrecen
  - Research Site, Pécs
  - Research Site, Szeged
  - Research Site, Székesfehérvár
  - Research Site, Tatabánya
  - Research Site, Zalaegerszeg
- Israel (7):
  - Research Site, Haifa
  - Research Site, Jerusalem
  - Research Site, Kfar Saba
  - Research Site, Petah Tikva
  - Research Site, Rehovot
  - Research Site, Rishon LeZiyyon
  - Research Site, Tel Aviv
- Italy (6):
  - Research Site, Bologna
  - Research Site, Florence
  - Research Site, Milan
  - Research Site, Roma
  - Research Site, Rozzano
  - Research Site, Udine
- Japan (20):
  - Research Site, Akita
  - Research Site, Amagasaki
  - Research Site, Asahikawa
  - Research Site, Chiyoda City
  - Research Site, Chūō
  - Research Site, Fukuoka
  - Research Site, Fukushima
  - Research Site, Hamamatsu
  - Research Site, Himeji
  - Research Site, Hirakata
  - Research Site, Kita-ku
  - Research Site, Kurume
  - Research Site, Meguro City
  - Research Site, Nagasaki
  - Research Site, Nagoya
  - Research Site, Sapporo
  - Research Site, Shinjuku-Ku
  - Research Site, Suita
  - Research Site, Toride
  - Research Site, Yokosuka
- Poland (7):
  - Research Site, Bielsko-Biala
  - Research Site, Bydgoszcz
  - Research Site, Krakow
  - Research Site, Lodz
  - Research Site, Olsztyn
  - Research Site, Tarnów
  - Research Site, Warsaw
- Russia (5):
  - Research Site, Chelyabinsk
  - Research Site, Kazan'
  - Research Site, Moscow
  - Research Site, Novosibirsk
  - Research Site, Saint Petersburg
- Ukraine (7):
  - Research Site, Kharkiv
  - Research Site, Kherson
  - Research Site, Kropyvnytskyi
  - Research Site, Lutsk
  - Research Site, Odesa
  - Research Site, Poltava
  - Research Site, Zaporizhzhya

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Balser S, Capsius B, Hole R, Papp A, Preissinger N, Rozenknop A, Tiko T. Randomised, double-masked trial to compare the efficacy, safety and immunogenicity of the biosimilar aflibercept FYB203 with reference aflibercept in patients with neovascular age-related macular degeneration. BMJ Open Ophthalmol. 2026 Jan 5;11(1):e002398. doi: 10.1136/bmjophth-2025-002398. PMID 41494750

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Only 1 eye was selected from each patient as the study eye. Patients with signs of nAMD in the fellow eye likely to require IVT anti-VEGF treatment during the study were excluded. Any necessary treatment for wAMD in the fellow eye was prohibited for the first eight weeks and could only occur with Eylea at least 14 days after study eye treatment, without classifying the fellow eye as a study eye.
Period: Overall Study
Arm/Group | FYB203 (Proposed Aflibercept Biosimilar) | Eylea® (Aflibercept)
Started | 215 | 219
Completed | 196 | 206
Not Completed | 19 | 13

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set (SAF)
Groups:
- Total: Total of all reporting groups
Arm/Group | FYB203 (Proposed Aflibercept Biosimilar) | Eylea® (Aflibercept) | Total
Number analyzed (Participants) | 215 | 218 | 433
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.7 (7.72) | 73.3 (7.70) | 73.5 (7.71)
Age, Customized [Count of Participants; unit: Participants]
  Age, Categorical: Between 18 and 64 years | 17 | 25 | 42
  Age, Categorical: Between 65 and 84 years | 181 | 180 | 361
  Age, Categorical: >= 85 years | 17 | 13 | 30
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 121 | 127 | 248
  Male | 94 | 91 | 185
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 5 | 8
  Not Hispanic or Latino | 212 | 213 | 425
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 17 | 16 | 33
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 197 | 201 | 398
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Bulgaria | 10 | 11 | 21
  Czechia | 34 | 35 | 69
  Hungary | 34 | 34 | 68
  Israel | 6 | 6 | 12
  Italy | 9 | 9 | 18
  Japan | 17 | 16 | 33
  Poland | 37 | 40 | 77
  Russia | 35 | 36 | 71
  Ukraine | 33 | 31 | 64

OUTCOME MEASURES:

1. Primary Outcome: Evaluate and Compare Functional Changes in Best Corrected Visual Acuity (BCVA) by Early Treatment Diabetic Retinopathy Study (ETDRS) Letters at Week 8 of Treatment With FYB203 or Eylea Compared to Baseline.
Description: Changes in Best Corrected Visual Acuity (BCVA) by ETDRS letters from the Baseline Visit (Visit 1) to Week 8 (Visit 3) were assessed. This involved measuring the number of letters a participant could correctly read using the study eye on the ETDRS chart. An increase in the number of ETDRS letters from baseline signifies an improvement in visual acuity of the study eye. The change from baseline was calculated as the observed post-baseline value minus the baseline value.
Time Frame: Week 8
Population: Full Analysis Set (FAS)
Measure: Least Squares Mean (Standard Error); unit: letters
Arm/Group | FYB203 (Proposed Aflibercept Biosimilar) | Eylea® (Aflibercept)
Number analyzed (Participants) | 215 | 218
letters | 6.6 (0.73) | 5.6 (0.73)
Statistical Analysis 1: Comparison: FYB203 (Proposed Aflibercept Biosimilar) vs Eylea® (Aflibercept); Test type: Equivalence — If the confidence interval for difference in LSMeans is completely contained in the interval ]-3.5 letters; 3.5 letters[, FBY203 and Eylea are considered equivalent; LS mean difference = 1.0, 90.4% CI 2-sided [-0.3 to 2.2], Standard Error of Mean 0.76

2. Secondary Outcome: Evaluate and Compare Functional Changes of the Retina by BCVA Over Time
Description: Change of BCVA by ETDRS letters over the whole study from Baseline Visit (Visit 1) to Week 24 (Visit 5) and Week 56 (Visit 9) - FAS
Time Frame: Through study completion, until Week 56 (Visit 9)
Population: FAS = Full Analysis Set
Measure: Mean (Standard Deviation); unit: letters
Arm/Group | FYB203 (Proposed Aflibercept Biosimilar) | Eylea® (Aflibercept)
Number analyzed (Participants) | 215 | 218
letters
  to Week 24 (Visit 5): number analyzed (Participants) | 201 | 203
  to Week 24 (Visit 5) | 7.0 (9.45) | 6.6 (9.51)
  to Week 56 (Visit 9): number analyzed (Participants) | 188 | 201
  to Week 56 (Visit 9) | 8.3 (10.37) | 6.6 (11.47)

3. Secondary Outcome: Evaluate and Compare Changes in Foveal Center Point (FCP) Retinal Thickness
Description: Change from Baseline Visit (Visit 1) in foveal center point FCP retinal thickness to Week 4 (Visit 2), Week 24 (Visit 5) and Week 56 (Visit 9) - FAS
Time Frame: Through study completion, until Week 56 (Visit 9)
Population: FAS = Full Analysis Set
Measure: Mean (Standard Deviation); unit: μm
Arm/Group | FYB203 (Proposed Aflibercept Biosimilar) | Eylea® (Aflibercept)
Number analyzed (Participants) | 215 | 218
μm
  to Week 4 (Visit 2): number analyzed (Participants) | 200 | 205
  to Week 4 (Visit 2) | -163.9 (142.17) | -168.4 (126.36)
  to Week 24 (Visit 5): number analyzed (Participants) | 186 | 189
  to Week 24 (Visit 5) | -165.9 (174.98) | -172.4 (153.00)
  to Week 56 (Visit 9): number analyzed (Participants) | 175 | 187
  to Week 56 (Visit 9) | -188.4 (181.08) | -202.4 (156.96)

4. Secondary Outcome: Evaluate and Compare the Proportion of Patients Who Gain or Lose ≥ 5, 10, and 15 Early Treatment Diabetic Retinopathy Study (ETDRS) Letters Compared to Baseline
Description: Proportion of patients who gain or lose ≥ 5, 10, or 15 Early Treatment Diabetic Retinopathy Study (ETDRS) letters from Baseline Visit (Visit 1) to Week 24 (Visit 5) and Week 56 (Visit 9) - FAS
Time Frame: Through study completion, until Week 56 (Week 9)
Population: FAS = Full Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | FYB203 (Proposed Aflibercept Biosimilar) | Eylea® (Aflibercept)
Number analyzed (Participants) | 215 | 218
Participants
  to Week 24 (Visit 5): number analyzed (Participants) | 201 | 203
  to Week 24 (Visit 5): ≥ 15 letters (gain 15 or more) | 45 | 38
  to Week 24 (Visit 5): ≥ 10 and < 15 letters (gain 10-14) | 41 | 39
  to Week 24 (Visit 5): ≥ 5 and < 10 letters (gain 5-9) | 41 | 47
  to Week 24 (Visit 5): > -5 and < 5 letters (gain or loss up to 4) | 52 | 58
  to Week 24 (Visit 5): > -10 and ≤ -5 letters (loss 5-9) | 12 | 13
  to Week 24 (Visit 5): > -15 and ≤ -10 letters (loss 10-14) | 6 | 2
  to Week 24 (Visit 5): ≤ -15 letters (loss 15 or more) | 4 | 6
  to Week 56 (Visit 9): number analyzed (Participants) | 188 | 201
  to Week 56 (Visit 9): ≥ 15 letters (gain 15 or more) | 52 | 49
  to Week 56 (Visit 9): ≥ 10 and < 15 letters (gain 10-14) | 43 | 36
  to Week 56 (Visit 9): ≥ 5 and < 10 letters (gain 5-9) | 34 | 39
  to Week 56 (Visit 9): > -5 and < 5 letters (gain or loss up to 4) | 39 | 48
  to Week 56 (Visit 9): > -10 and ≤ -5 letters (loss 5-9) | 12 | 13
  to Week 56 (Visit 9): > -15 and ≤ -10 letters (loss 10-14) | 6 | 7
  to Week 56 (Visit 9): ≤ -15 letters (loss 15 or more) | 2 | 9

5. Secondary Outcome: Evaluate and Compare the Absence of Disease Activity (Fluid-free Macula) Over Time
Description: Percentage of patients with fluid-free macula at Baseline (Visit 1), Week 24 (Visit 5), Week 56 (Visit 9) - FAS
Time Frame: Through study completion, until Week 56 (Visit 9)
Population: FAS = Full Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | FYB203 (Proposed Aflibercept Biosimilar) | Eylea® (Aflibercept)
Number analyzed (Participants) | 215 | 218
Participants
  Baseline (Visit 1): number analyzed (Participants) | 214 | 217
  Baseline (Visit 1): Assessment / Response = Yes | 0 | 0
  Baseline (Visit 1): Assessment / Response = No | 214 | 217
  Week 24 (Visit 5): number analyzed (Participants) | 198 | 200
  Week 24 (Visit 5): Assessment / Response = Yes | 71 | 65
  Week 24 (Visit 5): Assessment / Response = No | 127 | 135
  Week 56 (Visit 9): number analyzed (Participants) | 187 | 198
  Week 56 (Visit 9): Assessment / Response = Yes | 79 | 100
  Week 56 (Visit 9): Assessment / Response = No | 108 | 98

6. Secondary Outcome: Evaluate and Compare Systemic Free Aflibercept Concentrations in a Subgroup of up to 60 Patients (up to 30 Per Arm)
Description: Systemic concentrations (close to maximum concentration [Cmax]) of free aflibercept in a subgroup at selected sites - PKS:
  - 48 hours after the 3rd dose (Visit 3a)
Time Frame: At Baseline and Visit 3a (48 hours after the 3rd dose)
Population: PKS = Plasma Concentration Analysis Set. Baseline values that were reported as <LLOQ were analyzed with a numeric value of 0.5*LLOQ.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | FYB203 (Proposed Aflibercept Biosimilar) | Eylea® (Aflibercept)
Number analyzed (Participants) | 31 | 26
ng/mL
  Baseline (Visit 1): number analyzed (Participants) | 30 | 26
  Baseline (Visit 1) | 2.000 (0.0000) | 2.000 (0.0000)
  Visit 3a (48h after 3rd dose): number analyzed (Participants) | 31 | 25
  Visit 3a (48h after 3rd dose) | 122.166 (30.5161) | 120.112 (28.9556)

7. Secondary Outcome: Evaluate and Compare Change in Vision-related Functioning and Well-being Measured by National Eye Institute Visual Function Questionnaire 25 (NEI VFQ-25)
Description: Change from Baseline Visit (Visit 1) in vision-related functioning and well-being measured by National Eye Institute Visual Function Questionnaire 25 (NEI VFQ-25) to Week 24 (Visit 5) and Week 56 (Visit 9) - FAS. The NEI VFQ-25 includes 12 subscales (e.g., general vision, ocular pain, driving, peripheral vision) scored from 0 to 100, where higher scores indicate better functioning. Subscales are averaged to produce a composite score, excluding the general health subscale. Both subscale and composite scores range from 0 (worst) to 100 (best), representing the percentage of the highest possible score achieved.
Time Frame: Through study completion, until Week 56 (Visit 9)
Population: FAS = Full Analysis Set
Measure: Mean (Standard Deviation); unit: score points
Arm/Group | FYB203 (Proposed Aflibercept Biosimilar) | Eylea® (Aflibercept)
Number analyzed (Participants) | 215 | 218
score points
  to Week 24 (Visit 5): number analyzed (Participants) | 199 | 202
  to Week 24 (Visit 5) | 3.8 (11.06) | 1.8 (10.97)
  to Week 56 (Visit 9): number analyzed (Participants) | 190 | 201
  to Week 56 (Visit 9) | 3.8 (12.22) | 1.7 (12.46)

8. Secondary Outcome: Evaluate and Compare the Immunogenic Profile (Anti-drug Antibodies [ADAs]) in Serum
Description: Number of patients with anti-drug antibodies (ADAs) at Baseline (Visit 1), Week 24 (Visit 5) and Week 56 (Visit 9) - SAF
Time Frame: Through study completion, until Week 56 (Visit 9)
Population: SAF = Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | FYB203 (Proposed Aflibercept Biosimilar) | Eylea® (Aflibercept)
Number analyzed (Participants) | 215 | 218
Participants
  Week 1 (Baseline): number analyzed (Participants) | 213 | 204
  Week 1 (Baseline): Positive | 4 | 3
  Week 1 (Baseline): Negative | 209 | 201
  Week 24 (Visit 5): number analyzed (Participants) | 195 | 193
  Week 24 (Visit 5): Positive | 4 | 1
  Week 24 (Visit 5): Negative | 191 | 192
  Week 56 (Visit 9): number analyzed (Participants) | 194 | 192
  Week 56 (Visit 9): Positive | 5 | 2
  Week 56 (Visit 9): Negative | 189 | 190

9. Secondary Outcome: Frequency of Local and Systemic Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: Frequency of local and systemic adverse events (AEs) and serious adverse events (SAEs) - SAF
Time Frame: Through study completion, until Week 56 (Visit 9)
Population: SAF = Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | FYB203 (Proposed Aflibercept Biosimilar) | Eylea® (Aflibercept)
Number analyzed (Participants) | 215 | 218
Participants
  SAEs | 19 | 28
  local AEs, study eye | 67 | 75
  local AEs, fellow eye | 45 | 48
  systemic AEs | 124 | 113

ADVERSE EVENTS:
Time Frame: All AEs reported until the final end of study visit at week 56 are included.
Description: Safety analysis was performed on all patients who received at least 1 injection of study medication in the study eye. Patients were analyzed according to the treatment they actually received in the study eye irrespective of their randomized treatment.
Groups:
- FYB203 (Proposed Aflibercept Biosimilar), Systemic AE: Patients will receive intravitreal (IVT) injections of FYB203 as detailed in the protocol.
  FYB203 (Proposed aflibercept biosimilar): Patients will receive 1 IVT injection of FYB203 in the study eye only every 4 weeks for the first 3 consecutive doses, followed by 1 IVT injection every 8 weeks through study completion.
  In this column all systemic AEs by patient for the FYB203 group are given.
- Eylea® (Aflibercept), Systemic AE: Patients will receive intravitreal (IVT) injections of Eylea® as detailed in the protocol.
  Eylea® (Aflibercept): Patients will receive 1 IVT injection of Eylea® in the study eye only every 4 weeks for the first 3 consecutive doses, followed by 1 IVT injection every 8 weeks through study completion.
  In this column all systemic AEs by patient for the Eylea® group are given.
- FYB203 (Proposed Aflibercept Biosimilar), Ocular AE, Study Eye: Patients will receive intravitreal (IVT) injections of FYB203 as detailed in the protocol.
  FYB203 (Proposed aflibercept biosimilar): Patients will receive 1 IVT injection of FYB203 in the study eye only every 4 weeks for the first 3 consecutive doses, followed by 1 IVT injection every 8 weeks through study completion.
  In this column all ocular AEs by patient for the FYB203 group occurring in the study eye are given.
- Eylea® (Aflibercept), Ocular AE, Study Eye: Patients will receive intravitreal (IVT) injections of Eylea® as detailed in the protocol.
  Eylea® (Aflibercept): Patients will receive 1 IVT injection of Eylea® in the study eye only every 4 weeks for the first 3 consecutive doses, followed by 1 IVT injection every 8 weeks through study completion.
  In this column all ocular AEs by patient for the Eylea® group occurring in the study eye are given.
- FYB203 (Proposed Aflibercept Biosimilar), Ocular AE, Fellow Eye: Patients will receive intravitreal (IVT) injections of FYB203 as detailed in the protocol.
  FYB203 (Proposed aflibercept biosimilar): Patients will receive 1 IVT injection of FYB203 in the study eye only every 4 weeks for the first 3 consecutive doses, followed by 1 IVT injection every 8 weeks through study completion.
  The fellow eye could be treated with Eylea®, which was allowed after Visit 3 and was to be separated by at least 14 days from study eye treatment. In this group, 19 patients choose to get treatment for the fellow eye (from 1 to 6 injections).
  In this column all ocular AEs by patient for the FYB203 group occurring in the fellow eye are given.
- Eylea® (Aflibercept), Ocular AE, Fellow Eye: Patients will receive intravitreal (IVT) injections of Eylea® as detailed in the protocol.
  Eylea® (Aflibercept): Patients will receive 1 IVT injection of Eylea® in the study eye only every 4 weeks for the first 3 consecutive doses, followed by 1 IVT injection every 8 weeks through study completion.
  The fellow eye could be treated with Eylea®, which was allowed after Visit 3 and was to be separated by at least 14 days from study eye treatment. In this group, 20 patients choose to get treatment for the fellow eye (from 1 to 6 injections).
  In this column all ocular AEs by patient for the Eylea® group occurring in the fellow eye are given.
Arm/Group | FYB203 (Proposed Aflibercept Biosimilar), Systemic AE | Eylea® (Aflibercept), Systemic AE | FYB203 (Proposed Aflibercept Biosimilar), Ocular AE, Study Eye | Eylea® (Aflibercept), Ocular AE, Study Eye | FYB203 (Proposed Aflibercept Biosimilar), Ocular AE, Fellow Eye | Eylea® (Aflibercept), Ocular AE, Fellow Eye
All-Cause Mortality (participants affected / at risk) | 4/215 | 1/218 | 0/215 | 0/218 | 0/215 | 0/218
Serious Adverse Events (participants affected / at risk) | 17/215 | 23/218 | 2/215 | 2/218 | 0/215 | 3/218
Other Adverse Events (participants affected / at risk) | 56/215 | 46/218 | 44/215 | 49/218 | 37/215 | 32/218
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FYB203 (Proposed Aflibercept Biosimilar), Systemic AE (N=215) | Eylea® (Aflibercept), Systemic AE (N=218) | FYB203 (Proposed Aflibercept Biosimilar), Ocular AE, Study Eye (N=215) | Eylea® (Aflibercept), Ocular AE, Study Eye (N=218) | FYB203 (Proposed Aflibercept Biosimilar), Ocular AE, Fellow Eye (N=215) | Eylea® (Aflibercept), Ocular AE, Fellow Eye (N=218)
COVID-19 (Infections and infestations) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colonic abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Coronavirus infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gallbladder empyema (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peritonitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Toxic shock syndrome (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urosepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gallbladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oesophageal carcinoma stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Parathyroid tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Glaucoma (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Iridocyclitis (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neovascular age-related macular degeneration (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Retinal degeneration (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rhegmatogenous retinal detachment (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Uveitis (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Visual impairment (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal adhesions (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diverticulum intestinal (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Large intestinal stenosis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oesophageal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dementia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Transient global amnesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Clavicle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ligament injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nerve root injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diabetic metabolic decompensation (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Biliary dilatation (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gallbladder disorder (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aortic aneurysm (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Varicose vein (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Corneal dystrophy (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Calculus urinary (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FYB203 (Proposed Aflibercept Biosimilar), Systemic AE (N=215) | Eylea® (Aflibercept), Systemic AE (N=218) | FYB203 (Proposed Aflibercept Biosimilar), Ocular AE, Study Eye (N=215) | Eylea® (Aflibercept), Ocular AE, Study Eye (N=218) | FYB203 (Proposed Aflibercept Biosimilar), Ocular AE, Fellow Eye (N=215) | Eylea® (Aflibercept), Ocular AE, Fellow Eye (N=218)
Neovascular age-related macular degeneration (Eye disorders) | 0 (0) | 0 (0) | 7 (9) | 7 (9) | 22 (22) | 24 (25)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 8 (9) | 7 (7) | 7 (7) | 4 (4)
Conjunctival haemorrhage (Eye disorders) | 0 (0) | 0 (0) | 4 (4) | 14 (24) | 1 (1) | 0 (0)
Visual acuity reduced (Eye disorders) | 0 (0) | 0 (0) | 7 (7) | 4 (4) | 2 (2) | 2 (2)
Eye pain (Eye disorders) | 0 (0) | 0 (0) | 6 (6) | 6 (9) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 6 (6) | 3 (3) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 15 (17) | 17 (17) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 10 (11) | 6 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 5 (6) | 6 (6) | 5 (5) | 0 (0)
Coronavirus infection (Infections and infestations) | 5 (5) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 6 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 9 (10) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intraocular pressure increased (Investigations) | 0 (0) | 0 (0) | 7 (9) | 9 (25) | 2 (2) | 1 (1)
Hypertension (Vascular disorders) | 15 (16) | 9 (12) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 4 (4) | 7 (12) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2022-07-15): https://cdn.clinicaltrials.gov/large-docs/67/NCT04522167/Prot_000.pdf
  • Statistical Analysis Plan (2023-03-29): https://cdn.clinicaltrials.gov/large-docs/67/NCT04522167/SAP_001.pdf